CLINICAL TRIAL: NCT03001206
Title: The Use of Master Caution System for Continuous Monitoring and Detection of Dysrhythmia and Ischemia
Brief Title: The Use of the Master Caution System (MCS) for Continuous Monitoring and Detection of Dysrhythmias and Ischemic Events
Status: Completed | Type: Observational
Sponsor: HealthWatch Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-MCG-02
Record Dates: First submitted 2016-12-07; First posted 2016-12-22 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICCU patients: The use of the Master Caution System (MCS) for continuous monitoring and detection of dysrhythmias and ischemic events :
  For patient diagnosed with acute coronary syndrome (ACS) in the intensive cardiac care unit (ICCU) before and after planed catheterization procedure.
  Interventions: Device: Master Caution System
- Stress test subjects: The use of the Master Caution System (MCS) for continuous monitoring and detection of dysrhythmias and ischemic events :
  For patients referred to stress imaging with suspected ischemia.
  Interventions: Device: Master Caution System

INTERVENTIONS:
Device: Master Caution System — The purpose of this study is to evaluate the effectiveness and usability of the Master Caution System for 12 leads continuous monitoring of ECG signal in the ICCU.
  The purpose of the study is to evaluate the effectiveness and usability of using Master Caution 12 leads Garment for stress test.
  The purpose of the study is to reassess the adequate size of the Master Caution Garment (MCG).

SUMMARY:
The purpose of this study is to evaluate the effectiveness and usability of the Master Caution System for 12 leads continuous monitoring of ECG signal in the ICCU.

The purpose of the study is to evaluate the effectiveness and usability of using Master Caution 12 leads Garment for stress test.

The purpose of the study is to reassess the adequate size of the Master Caution Garment.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Diagnosed or have evidence of ACS, or referred for stress imaging due to suspected ischemia with STT changes.
* Needs continuous/routine ECG monitoring.
* Ability to give informed consent.
* Cooperative person

Exclusion Criteria:

* Patients with known allergy to silver.
* Patients with dermal disease or recent trauma to the chest wall.
* Pregnant or lactating woman.
* Patients with chest deformity precluding placement of the garment.
* Patients suffering from tremor.
* Patients participating in another ongoing trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects admitted and diagnosed as acute coronary syndrome, before or after catheterization, who need to be monitored for evaluation of treatment efficacy.
  Eligible subjects referred to stress imaging test, with current or previously depicted STT changes.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Measuring 12 leads ECG information of patients at the ICCU in continuous monitoring using Master Caution System (MCS) will give more cardiac information comparing to regular hospital 2-3 leads telemetry. | 48 hours
Measuring 12 leads ECG information of patients at the stress test using Master Caution System (MCS) comparing to the standard of care stress test ECG device and Electrodes. | 1-2 hours

SECONDARY OUTCOMES:
Master Caution System (MCS) cardiac telemetry system will measure and provide sufficient ECG information for adequate detection and interpretation of ST-T wave changes and dysrhythmic events. | during the use of the system

CONTACTS AND LOCATIONS:
Overall Officials: Morris Mosseri, Prof., Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No